CLINICAL TRIAL: NCT01889797
Title: Phase II Randomized Trial Comparing GA101 (Obinutuzumab) and Rituximab in Patients With Previously Untreated Low Tumor Burden Indolent Non-Hodgkin's Lymphoma
Brief Title: Phase II Randomized Trial Comparing GA101 and Rituximab in Untreated Low Tumor Burden Indolent Non-Hodgkin's Lymphoma
Acronym: PrE0401
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due prolonged enrollment timelines
Sponsor: PrECOG, LLC. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrE0401; BO25454 (Other Grant/Funding Number: Genentech)
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Indolent Non-Hodgkin's Lymphoma
Keywords: Untreated Non-Hodgkin's Lymphoma; Low Tumor Burden Non-Hodgkin's Lymphoma; NHL; Indolent; Rituximab; Rituxan; GA101; Obinutuzumab
MeSH Terms: interventions — Rituximab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Rituximab (Active Comparator): Rituximab 375 mg/m² IV weekly for 4 weeks.
  Interventions: Biological: Arm A: Rituximab
- Arm B: GA101 (Experimental): GA101 1,000 mg IV weekly for 4 weeks.
  Interventions: Biological: Arm B: GA101

INTERVENTIONS:
Biological: Arm A: Rituximab — Rituximab 375 mg/m² IV x 4 weekly doses.
  Other Names: IDEC-C2B8; Chimeric anti-CD20 monoclonal antibody; Rituxan; NSC# 687451
  Arms: Arm A: Rituximab
Biological: Arm B: GA101 — GA101 1,000 mg (flat dose) IV x 4 weekly doses.
  Other Names: Obinutuzumab; RO5072759; huMAB<CD20>
  Arms: Arm B: GA101

SUMMARY:
Patients with previously untreated low tumor burden indolent Non-Hodgkin's Lymphoma (NHL) will receive either rituximab or GA101 weekly for 4 weeks followed by re-staging to determine response.

Rituximab, an anti-CD20 chimeric antibody, was approved by the United States Food and Drug Administration in 1998 for the treatment of patients with relapsed low-grade B-cell lymphomas. Clinically, four weekly doses of rituximab have proven to be well tolerated and effective in previously untreated as well as relapsed patients with low-grade lymphoma.

GA101 is an anti-CD20 humanized and glyco-engineered monoclonal antibody. GA101 has been shown to have increased antibody-dependent cellular cytotoxicity (ADCC) and direct cell-death induction compared to Rituximab. It is possible that GA101 may have greater efficacy than rituximab.

PrE0401 Sub-Study Evaluation of Corrected QT (QTc) Interval and Pharmacokinetic Parameters in Patients Participating in GA101 (Obinutuzumab)

Approximately twenty-five patients randomized to GA101 may participate in the sub-study. Electrocardiograms and blood samples will be obtained.

DETAILED DESCRIPTION:
According to the American Cancer Society, it is estimated that approximately 70,800 individuals will be diagnosed with non-Hodgkin's lymphoma (NHL) and over 18,990 men and women will die of the disease in 2014. The survival rates for patients with indolent NHL remained unchanged from the 1950s through the early 1990s, but recent evidence suggests that outcomes are improving. Indolent NHL is a particular challenge because it is an incurable disease requiring multiple treatments; yet relatively long survivals elevate the importance of quality of life associated with treatment.

Agents such as rituximab are active in patients with a low burden of disease and result in high response rates and durable remissions for most patients. However, the optimal therapeutic approach to patients with low-grade lymphoma with a low disease burden is controversial as conventional chemotherapy also results in high rates of response. Regardless of whether patients receive immunotherapy, chemotherapy, or a combination thereof, they unfortunately exhibit a continuing pattern of disease relapse and the median survival for newly diagnosed patients is between 7-10 years.

Rituximab and GA101 both target the CD20 antigen. The CD20 antigen is located on the surface of normal and malignant B-cell lymphocytes. An attractive feature of this target is that CD20 is not on hematopoietic stem cells, nor is it expressed in any great extent on other normal body tissues.

Studies in vitro have shown that rituximab predominantly induces antibody dependent cellular cytotoxicity (ADCC), but also binds complement and directly induces apoptosis in lymphoma cells.

GA101 shows increased ADCC related to an improved binding of the GA101 to the different allotypes expressed by natural killer cells and monocytes. It also has increased direct cell-death related to an elbow hinge amino acid exchange and Type II binding of the CD20 epitope. The safety of GA101 in NHL so far appears to be similar to that observed with rituximab in patients with NHL, except for a higher incidence of infusion-related reactions.

Depletion of malignant B-cells using anti-CD20 monoclonal antibodies has an acceptable safety profile, particularly in patients with low-grade B-cell lymphomas with a low disease burden. To determine whether treatment with GA101 results in better outcomes than that seen with rituximab and to determine which anti-CD20 antibody to utilize in future studies, we will conduct a randomized Phase II trial of rituximab and GA101 in patients with previously untreated low-grade lymphoma. Patients will receive either rituximab or GA101 weekly for 4 weeks followed by re-staging. The endpoints of the study will be the Complete Response (CR), Overall Response Rate (ORR), time to next treatment, progression free survival (PFS), and safety of each treatment arm.

PrE0401 Sub-Study Evaluation of Corrected QT (QTc) Interval and Pharmacokinetic Parameters in Patients Participating in GA101 (Obinutuzumab)

Patients randomized to GA101 and who consent to the sub-study will have electrocardiograms obtained pre and post Week 1 and Week 4 to investigate the effect of GA101 on QTc interval. Pharmacokinetic blood samples will also be done to evaluate serum concentrations of GA101 at the same time-points.

ELIGIBILITY:
Inclusion Criteria:

Registration: Patients having both diffuse and follicular architectural elements will be considered eligible if the histology is predominantly follicular (≥ 50% of the cross-sectional area), and there is no evidence of transformation to a large cell histology.

* Biopsy-proven diagnosis of Grade 1 or 2 follicular non-Hodgkin's lymphoma with no evidence of transformation to large cell histology.
* Meet criteria for Low Tumor Burden:

  * No nodal or extra nodal mass ≥ 7 centimeter (cm)
  * <3 nodal masses >3 cm in diameter
  * No systemic symptoms or B symptoms
  * No splenomegaly >16 cm by CT scan
  * No risk of compression of a vital organ.
  * No leukemic phase with >5000/mm³ circulating lymphocytes.
* No cytopenias defined as:

  * Platelets <100,000/mm³
  * Hemoglobin (Hgb) <10 g/dL
  * Absolute Neutrophil Count (ANC) <1500/mm³
* Must have Stage III or Stage IV disease.
* Baseline measurements/evaluations obtained within 6 weeks of registration. Patient must have at least one objective measurable disease parameter.
* Age ≥ 18 years.
* Eastern Oncology Cooperative Group Performance Status 0-1.
* Must not have received investigational agents within 30 days of registration.
* Signed Institutional Review Board (IRB)-approved informed consent.
* Willing to provide blood samples for research purposes.
* Women must not be pregnant or breastfeeding.
* Women of childbearing potential and sexually active males must use an accepted and effective method of contraception.
* No prior chemotherapy, radiotherapy or immunotherapy for lymphoma.
* No prior treatment with cytotoxic drugs or rituximab for a previous cancer or another condition (e.g. rheumatoid arthritis) or prior use of an anti-CD20 antibody.
* No prior use of any monoclonal antibody within 3 months of randomization.
* No history of severe allergic/anaphylactic reactions to humanized/murine monoclonal antibodies or known sensitivity/allergy to murine products.
* No history of prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least 2 years and did not require treatment with cytotoxic drugs or rituximab.
* No major surgery within 4 weeks prior to randomization, other than for diagnosis.
* Must be Human Immunodeficiency Virus (HIV) negative.
* Have adequate organ function without growth factor and/or transfusion support within ≤ 2 weeks prior to registration:

  * ANC ≥ 1500/mm³
  * Hgb ≥ 10 g/dL
  * Platelets ≥ 100,000/mm³
  * Serum Creatinine ≤ 2x Upper Limit Normal (ULN)
  * Total Bilirubin ≤ 2x ULN
  * AST (aspartate aminotransferase)/ALT (alanine aminotransferase) ≤ 5x ULN
  * PTT (Partial Thromboplastin Time) or aPTT (activated Partial Thromboplastin Time) >1.5x the ULN in the absence of a lupus anticoagulant
  * INR (International Normalized Ratio) >1.5x the ULN in the absence of therapeutic anticoagulation
* No active, uncontrolled infections (afebrile for ≥ 48 hours off antibiotics).
* Must not receive immunization with attenuated live vaccines within 28 days prior to registration or during the study period.
* Must be tested for hepatitis B surface antigen (HBsAg) and total hepatitis B core antibody (anti-HBc) within 2 weeks of registration. Patients who are chronic carriers of HBsAg and anti-HBc are excluded.
* Must be tested for hepatitis C antibody within 2 week of registration. If this test is positive, patients are excluded unless a hepatitis C virus ribonucleic acid (HCV RNA) is negative.
* No evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (i.e., severe arrhythmia, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ansell, MD, Study Chair — Mayo Clinic in Minnesota
Locations (28):
- United States (28):
  - University of South Alabama, Mobile, Alabama
  - Marin Cancer Care, Greenbrae, California
  - St. Joseph's/Candler Health System, Savannah, Georgia
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University, Indianapolis, Indiana
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - St. Joseph Mercy Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro MN CCOP, Saint Louis Park, Minnesota
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Aultman Hospital, Canton, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Toledo Community Oncology Program, Toledo, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Susquehanna Health Cancer Center, Williamsport, Pennsylvania
  - University of Virginia, Charlottesburg, Virginia
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia
  - Gundersen Health System, La Crosse, Wisconsin
  - Dean Clinic, Madison, Wisconsin
  - ProHealth Care, Inc., Waukesha, Wisconsin
  - Aurora Health Care, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

REFERENCES:
- [Background] Hainsworth JD, Litchy S, Burris HA 3rd, Scullin DC Jr, Corso SW, Yardley DA, Morrissey L, Greco FA. Rituximab as first-line and maintenance therapy for patients with indolent non-hodgkin's lymphoma. J Clin Oncol. 2002 Oct 15;20(20):4261-7. doi: 10.1200/JCO.2002.08.674. PMID 12377971
- [Background] Beers SA, Chan CH, French RR, Cragg MS, Glennie MJ. CD20 as a target for therapeutic type I and II monoclonal antibodies. Semin Hematol. 2010 Apr;47(2):107-14. doi: 10.1053/j.seminhematol.2010.01.001. PMID 20350657
- [Background] Mossner E, Brunker P, Moser S, Puntener U, Schmidt C, Herter S, Grau R, Gerdes C, Nopora A, van Puijenbroek E, Ferrara C, Sondermann P, Jager C, Strein P, Fertig G, Friess T, Schull C, Bauer S, Dal Porto J, Del Nagro C, Dabbagh K, Dyer MJ, Poppema S, Klein C, Umana P. Increasing the efficacy of CD20 antibody therapy through the engineering of a new type II anti-CD20 antibody with enhanced direct and immune effector cell-mediated B-cell cytotoxicity. Blood. 2010 Jun 3;115(22):4393-402. doi: 10.1182/blood-2009-06-225979. Epub 2010 Mar 1. PMID 20194898
- [Background] Salles GA, et al. Efficacy and Safety of Obinutuzumab (GA101) Monotherapy in Relapsed/Refractory Indolent Non-Hodgkin's Lymphoma: Results from a Phase I/II Study (BO20999) American Society of Hematology Annual meeting 2011 Abstract 268.
- [Background] Sehn LH, Goy A, Offner FC, Martinelli G, Caballero MD, Gadeberg O, Baetz T, Zelenetz AD, Gaidano G, Fayad LE, Buckstein R, Friedberg JW, Crump M, Jaksic B, Zinzani PL, Padmanabhan Iyer S, Sahin D, Chai A, Fingerle-Rowson G, Press OW. Randomized Phase II Trial Comparing Obinutuzumab (GA101) With Rituximab in Patients With Relapsed CD20+ Indolent B-Cell Non-Hodgkin Lymphoma: Final Analysis of the GAUSS Study. J Clin Oncol. 2015 Oct 20;33(30):3467-74. doi: 10.1200/JCO.2014.59.2139. Epub 2015 Aug 17. PMID 26282650

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Rituximab | Arm B: GA101
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Rituximab | Arm B: GA101 | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Median (Full Range); unit: years] | 52 [37 to 81] | 59 [31 to 82] | 56 [31 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 6 | 11 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 16 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
ECOG Performance Status [Number; unit: participants] — The ECOG performance status (PS) measures how a disease impacts a patient's daily living abilities. It describes a patient's level of functioning in terms of their ability to care for themselves, daily & physical abilities. The PS score ranges from 0 to 5. A PS score of 0 indicates that a patient is fully active & able to carry out all pre-disease performance without restriction; 1 indicates that a patient is restricted in performance; 2 indicates ambulatory; & at the extreme, 5 indicates a patient is deceased. High score indicates the disease has a higher negative impact on living abilities.
  participants
    PS 0 | 12 | 12 | 24
    PS 1 | 4 | 4 | 8
Modified Ann Arbor Staging [Number; unit: participants] — The Ann Arbor staging is used to describe the extent of non-Hodgkin lymphoma (NHL) in adults. There are 4 levels of the Ann Arbor staging system. Stage I means the lymphoma is only in 1 lymph node area or lymphoid organ; II indicates 2 or more groups of lymph nodes on the same side of the diaphragm; III indicates disease is present in lymph node areas on both sides of the diaphragm and may have spread to other organs; and IV shows that disease has spread outside the lymph system and also to the bone marrow, liver, brain, spinal cord or lungs. Higher grades are considered as worse.
  participants
    Stage III (1) | 1 | 5 | 6
    Stage III (2) | 5 | 4 | 9
    Stage IV | 10 | 7 | 17
Primary Tumor Type [Number; unit: participants]
  Grade 1 Follicular NHL | 10 | 13 | 23
  Grade 2 Follicular NHL | 4 | 3 | 7
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate
Description: Positron Emission Tomography (PET)-documented CR rates after induction therapy (weekly treatment x 4 weeks with GA101 or rituximab)
  Definitions for clinical response are modified from the Revised Response Criteria for Malignant Lymphoma (Cheson BD, et al. Revised Response Criteria for Malignant Lymphoma. J Clin Oncol 2007; 25(5): 579-86). Lymph node measurements were taken from CT, CT portion of the PET/CT, or MRI scans where applicable. CR is defined as complete disappearance of all evidence of disease; PR as a >50% decrease in the sum of the products of the maximal perpendicular diameters of measured lesions (SPD) and no new sites; SD as failure to attain CR/PR or PD; and PD as any new lesion >1.5cm in any axis or ≥50% increase in previously involved sites.
Time Frame: Re-staging (week 12, 13 or 14) and during follow-up if physician feels patient is subsequently in CR for up to 4 years
Population: All participants were included in the analysis
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Rituximab | Arm B: GA101
Number analyzed (Participants) | 16 | 16
percentage of participants | 37.5 [21.0 to 56.5] | 56.2 [37.5 to 73.7]

2. Secondary Outcome: PET Response Rate
Description: PET response rate [PET-documented CR + Partial Response (PR)] based on PET scan results. Patients with unevaluable disease were included in the denominator.
Time Frame: Re-staging (week 12, 13 or 14)
Measure: Number; unit: participants
Arm/Group | Arm A: Rituximab | Arm B: GA101
Number analyzed (Participants) | 16 | 16
participants
  Complete Response | 6 | 9
  Partial Response | 5 | 5
  Stable Disease | 3 | 2
  Progressive Disease | 2 | 0

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate (CR + PR by Cheson criteria) at re-staging (including bone marrow biopsy if CR suspected) by PET and Neck, Chest, Abdomen and Pelvic Computed Tomography (CT) scan. Patients with unevaluable disease were included in the denominator.
Time Frame: Baseline and Re-staging (week 12, 13 or 14)
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Rituximab | Arm B: GA101
Number analyzed (Participants) | 16 | 16
percentage of participants | 68.8 [49.6 to 83.9] | 87.5 [70.0 to 96.6]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: CT scan every 3 months for 2 years, then every 6 months until progression. Compare PFS in each treatment arm.
  Progressive disease (PD) was defined using Cheson criteria as described in the Primary Outcome section above. Progression-free survival (PFS) was defined as the time from start of treatment to the documentation of PD or death, whichever occurs first. Patients alive and without PD were censored at the date of last disease assessment.
Time Frame: Percent of participants alive and progression-free at 1 year
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Rituximab | Arm B: GA101
Number analyzed (Participants) | 16 | 16
percentage of participants | 68.8 [44.2 to 84.2] | 87.5 [61.8 to 96.4]

ADVERSE EVENTS:
Description: Adverse events were assessed weekly, prior to and during administration of study drug.
Arm/Group | Arm A: Rituximab | Arm B: GA101
Serious Adverse Events (participants affected / at risk) | 0/16 | 2/16
Other Adverse Events (participants affected / at risk) | 11/16 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Rituximab (N=16) | Arm B: GA101 (N=16)
Flushing (Vascular disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Infusion Related Reaction (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Rituximab (N=16) | Arm B: GA101 (N=16)
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anxiety (Nervous system disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Asthenia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Alkaline Phosphatase Increased (Investigations) | 1 | 0
Chills (General disorders) | 1 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cytokine Release Syndrome (Immune system disorders) | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2
Dermatitis Allergic (Immune system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Edema (General disorders) | 1 | 0
Infusion Site Extravasation (General disorders) | 1 | 1
Eye Disorder (Eye disorders) | 0 | 1
Fatigue (General disorders) | 3 | 8
Headache (Nervous system disorders) | 1 | 3
Hot Flashes (Vascular disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Flu Like Symptoms (General disorders) | 0 | 1
Infusion Related Reaction (General disorders) | 5 | 6
Insomnia (Psychiatric disorders) | 0 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 4 | 3
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 2
Fever (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Blurred Vision (Eye disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study closed early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No